CLINICAL TRIAL: NCT04350476
Title: Remote Monitoring in Patients With Coronavirus Disease (COVID-19)
Brief Title: COVID-19 Remote Monitoring
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: closed due to lack of interest and enrollment
Sponsor: Vivek Reddy (Other)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GCO 20-0932
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: COVID-19; Cardiac Arrhythmias
Keywords: COVID-19; Cardiac Arrhythmias; Atrial Fibrillation; Telemetry
MeSH Terms: conditions — COVID-19; Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a non-randomized study. Based on clinical assessment, patients will be provided with the following home monitoring system: VitalConnect Vital Sign Patch (San Jose, California) This patch provides continuous real-time monitoring of cardiac telemetry, heart rate, respiratory rate and oxygen saturation. Duration of monitoring is typically up to 7 days.
  This patch is applied to the upper left side of the chest wall, attached with a hypoallergenic adhesive material. (This device is FDA approved for this indication).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Vital Connect Patch Arm (Other): This is a non-randomized study. Based on clinical assessment, patients will be provided with the following home monitoring system:
  VitalConnect Vital Sign Patch (FDA approved for this indication)
  Interventions: Diagnostic Test: VitalConnect Vital Sign Patch

INTERVENTIONS:
Diagnostic Test: VitalConnect Vital Sign Patch — This patch provides continuous real-time monitoring of cardiac telemetry, heart rate, respiratory rate and oxygen saturation. Duration of monitoring is typically up to 7 days.
  This patch is applied to the upper left side of the chest wall, attached with a hypoallergenic adhesive material. (This device is FDA approved for this indication).

SUMMARY:
The objective of the study is to assess the impact of remote cardiac and vital sign monitoring in patients with coronavirus disease (COVID-19) in the outpatient setting.

DETAILED DESCRIPTION:
The objective of the study is to assess the impact of remote cardiac and vital sign monitoring in patients with coronavirus disease (COVID-19) in the outpatient setting. This study will enroll COVID-19 positive patients previously evaluated at Mount Sinai Hospital/Mount Sinai Health System (MSHS) and affiliated hospitals deemed appropriate for home monitoring. Patients will be monitored remotely in the outpatient setting for 1-3 weeks following diagnosis and/or treatment for COVID-19 at MSH/MSHS.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with coronavirus and determined to be eligible for home monitoring and self-care, and either

  1. Not admitted to the hospital, and permitted to recover at home
  2. Discharged from inpatient hospitalization, during the acute recovery period
* 18 years old or older with the ability to understand the requirements of the study and sign the informed consent form (or able to provide over-the-phone verbal consent).

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Number of different arrhythmias | 7-14 Days
  ac rhythm in patients with COVID-19 infection following treatment/discharge from MSH
Temperature | 7-14 Days
  Temperature of patients with COVID-19 infection following treatment/discharge from MHS
Oxygen Saturation | 7-14 Days
  Oxygen saturation level in patients with COVID-19 infection following treatment/discharge from MSH

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Y Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Martin Goldman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai

IPD SHARING:
Plan to Share IPD: No